CLINICAL TRIAL: NCT05312814
Title: Clinical Utility of the Addition of a SNP-based NIPT Zygosity Determination in Twin Pregnancy Management.
Acronym: ZTWINS
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-051-NPT
Record Dates: First submitted 2022-02-24; First posted 2022-04-06 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Twin to Twin Transfusion Syndrome; Pregnancy Complications; Multiple Gestation; Maternal Care
MeSH Terms: conditions — Fetofetal Transfusion; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Twin pregnancies undergoing non-invasive prenatal screening: Women carrying a twin pregnancy undergoing non-invasive prenatal screening for zygosity and aneuploidy syndromes.
  No drug/device will be administered; clinical data will be collected for research analysis.

SUMMARY:
The ZTWINS registry study is an observational, prospective, multi-center study observing women carrying a twin pregnancy who receive snp-based non-invasive prenatal screening and zygosity assessment as part of their medical care.

DETAILED DESCRIPTION:
This observational data collection study will include subjects with ultrasound-confirmed twin pregnancy and planned NIPS zygosity assessment as a part of their clinical care. Initial chorionicity assessment and, when available, planned twin pregnancy management (e.g., frequency of prenatal ultrasounds, maternal fetal medicine (MFM) referral etc) will be recorded in the study database. Following zygosity results being returned through clinical care NIPS, updated chorionicity & amnionicity will again be recorded in the study database. Other clinical data in the medical record as part of clinical care, including monochorionic twin pregnancy complications (TTTS, FTC referral, etc), placenta pathology findings, and delivery and neonatal outcomes will also be recorded in the study database. There will be no study blood sample collection or other study procedures performed as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Women with an ultrasound confirmation of twin pregnancy

Exclusion Criteria:

* Singleton or non-twin multiple pregnancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women carrying a twin pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Assess clinical utility of combining NIPT-based zygosity measurements with ultrasound chorionicity assessments for the management of twin pregnancies. | 2 years
  Primary outcome will be measured by determining the overall frequency of NIPT-determined monozygosity among twin pregnancies; the frequency of discordance between NIPT-determined zygosity and ultrasound only chorionicity assessments; and the proportion of twin pregnancies with twin--twin transfusion syndrome (TTTS) that are diagnosed late as compared with historical rates.
Frequency of monozygosity | 2 years
  Measuring overall frequency of NIPT-determined monozygosity among twin pregnancies, measured by the number monozygotic pregnancies over the total number of twin pregnancies in the study.
Frequency of changed chorionicity assessment | 2 years
  The frequency of discordance between NIPT-determined zygosity and ultrasound only chorionicity assessments, as measured by the total number of pregnancies with a change in chorinicity assessment following the NIPT-based zygsity results release.
Frequency of late TTTS diagnosis | 2 years
  The frequency of late diagnosis of Twin to Twin Transfusion Syndrome (TTTS) in twin pregnancies with TTTS will be compared with historical rates of late TTTS diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Quintero, MD, Principal Investigator — The Fetal Institute
Locations (8):
- United States (8):
  - Rady Children Specialists of San Diego, San Diego Perinatal Center, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Anne Arundel Medical Center/Luminis Health, Annapolis, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Carnegie Imaging for Women, New York, New York
  - University of Rochester, Rochester, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Seven Hills/ Axia, Cincinnati, Ohio